CLINICAL TRIAL: NCT03831633
Title: A Pragmatic Randomized Study to Evaluate the Comparative Effectiveness of AKYNZEO® and Standard of Care (Including EMEND®) for the Prevention of Nausea and Vomiting (CINV) in Cancer Patients Receiving Moderately Emetogenic Chemotherapy in France.
Brief Title: Comparative Effectiveness of AKYNZEO® and Standard of Care (Including EMEND®) for the Prevention of Nausea and Vomiting (CINV) in Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRAKYFRA-01
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — netupitant, palosentron drug combination; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AKYNZEO (Experimental)
  Interventions: Drug: Akynzeo
- Standard of Care (Active Comparator)
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Akynzeo — 1 single oral dose of NEPA (capsule) on Day 1 to be administered approximately 1 hour prior chemotherapy (containing 300 mg netupitant and 0.5 mg palonosetron).
  - Dexamethasone 12 mg on Day 1 and 8 mg daily from Day 2 to Day 4
  Arms: AKYNZEO
Drug: Standard of Care — * oral aprepitant 125mg (Day 1) and 80mg daily (on Day 2 and Day 3)
  * IV ondansetron 8 mg on Day 1
  * Dexamethasone 12 mg on Day 1 and 8 mg daily from Day 2 to Day 4
  Arms: Standard of Care

SUMMARY:
This pragmatic trial addresses the clinical gap through the generation of evidence on the comparative effectiveness between AKYNZEO® and Standard of Care (SoC, including EMEND®) in the real-life setting

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Age ≥ 18 years
* Have a histological or cytological confirmed solid tumor malignancy
* Patient scheduled to receive their first course of anthracycline cyclophosphamide (AC) based chemotherapy regimen or Moderately Emetogenic Chemotherapy for the treatment of solid malignant tumor
* Patient scheduled to receive CINV prevention with AKYNZEO® or Standard of Care according to the summary of product characteristics based on the judgement of their investigator's
* Naïve of CT
* ECOG performance up to 2
* Able to read, understand and follow the study procedures
* Patient with Health insurance

Exclusion Criteria:

* Pregnancy and breastfeeding women;
* Hypersensitivity to active substances, excipients or other ingredients of Akynzeo® or Emend®;
* Protected patients: majors under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Anti-emetic response | 1 cycle (cycle length is 28 days). Primary outcome will be assessed at the end of the chemotherapy cycle.
  Complete Response (no emetic episodes and no rescue medication) during overall phase for 1st cycle among patients with MEC non AC or AC chemotherapy regimen

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Avicenne, Paris, France

IPD SHARING:
Plan to Share IPD: No